CLINICAL TRIAL: NCT07404891
Title: Single-Center, Randomized, Double-Blind, Parallel-Controlled Clinical Trial to Evaluate the Efficacy and Safety of ALT001 for Osteoarthritis
Brief Title: Clinical Trial on the Efficacy and Safety of ALT001 in Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALT001-CN-IIT-09002
Record Dates: First submitted 2026-02-04; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Group (Placebo Comparator): 2 vials per administration, once every 2 weeks, intra-articular injection.
  Interventions: Other: Placebo
- ALT001 Low-Dose Group (Experimental): 1 vial per administration, once every 2 weeks, intra-articular injection.
  Interventions: Drug: ALT001
- ALT001 High-Dose Group (Experimental): 2 vials per administration, once every 2 weeks, intra-articular injection.
  Interventions: Drug: ALT001

INTERVENTIONS:
Other: Placebo — Administration Method: Intra-articular injection; the medial and lateral joint spaces are recommended as the injection sites.
  Total Number of Injections: 6 times
  Arms: Placebo Group
Drug: ALT001 — Administration Method: Intra-articular injection; the medial and lateral joint spaces are recommended as the injection sites.
  Total Number of Injections: 6 times
  Arms: ALT001 High-Dose Group; ALT001 Low-Dose Group

SUMMARY:
This clinical trial will focus on the core efficacy endpoints including relief of pain intensity, improvement of joint motor function and enhancement of quality of life in patients. Meanwhile, it will strictly monitor key safety indicators such as the occurrence of various adverse events after medication, the severity and duration of adverse reactions, and conduct a multi-dimensional and multi-level comprehensive assessment. The study aims to clarify the clinical benefit profile and safety risks of the investigational product ALT001, and provide scientific, detailed and reliable evidence-based medical data to support the optimization of clinical treatment guidelines and the formulation of individualized treatment regimens for knee osteoarthritis.

Patients enrolled in the trial will receive investigational product treatment on the basis of conventional therapy. They will be randomly assigned to the placebo group, low-dose group and high-dose group at a ratio of 1:1:1. For each treatment course, patients in all groups will receive an injection of 2 vials of the investigational product into a single knee joint (for bilateral knee osteoarthritis, both knees may be injected, with one fixed knee joint selected for subsequent assessments). The injection will be administered once every 2 weeks for a total of 6 administrations.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled clinical trial. Patients will be enrolled after signing the informed consent form and meeting the inclusion/exclusion criteria, with a planned enrollment of 30 participants.

All enrolled patients will receive the study drug on the basis of conventional treatment, and be randomly assigned to the placebo group, low-dose group and high-dose group at a ratio of 1:1:1 (see Table 1 for details). Patients in each group will receive an injection of 2 vials of the study product into a single knee joint per treatment session (for bilateral osteoarthritis, both knees may be injected, while a fixed knee joint will be selected for subsequent assessments). Injections will be administered once every 2 weeks for a total of 6 times.

Follow-up assessments will be conducted concomitantly with injections at 2, 4, 6, 8 and 10 weeks after the first injection, and all safety and efficacy data will be collected during these visits.

The entire study consists of the following phases: Screening Period (Day -7 to Day 0), Treatment Visit 1 (first injection, Day 0), Treatment Visit 2 (second injection, Week 2 ±3 days), Treatment Visit 3 (third injection, Week 4 ±3 days), Treatment Visit 4 (fourth injection, Week 6 ±3 days), Treatment Visit 5 (fifth injection, Week 8 ±3 days), Treatment Visit 6 (sixth injection, Week 10 ±3 days), Follow-up Visit 7 (Week 12 ±5 days), Follow-up Visit 8 (Week 18 ±7 days) and Follow-up Visit 9 (Week 24 ±7 days).

The outcome measures of this clinical trial are based on the participants' subjective evaluations. To avoid bias in trial results caused by participants' subjective perceptions, a blinded design is applied to all participants. A double-blind design is also adopted, with follow-up investigators masked, to prevent the investigators' subjective judgments from influencing participants during follow-up. This trial uses a placebo-controlled design, where the trial conditions, clinical observation items and evaluation criteria are consistent between the experimental and control groups. In addition, participants in the two groups are assigned in accordance with the randomization principle.

This clinical trial is developed in response to the urgent clinical need for safe and effective interventions in the treatment of knee osteoarthritis. In accordance with the principles of evidence-based medicine, a rigorous controlled study protocol has been designed. Through standardized trial procedures and a unified evaluation system, this trial will systematically and comprehensively assess the clinical application value of ALT001, manufactured by Darwin Starting Point (Hubei) Biopharmaceutical Co., Ltd., in patients with knee osteoarthritis. The study will focus on core efficacy endpoints including the degree of pain relief, improvement in joint motor function and enhancement of quality of life in patients. Meanwhile, key safety indicators such as the incidence of various adverse events after administration, the severity and duration of adverse reactions will be closely monitored. A multi-dimensional and multi-level comprehensive assessment will be conducted to clarify the clinical benefit characteristics and safety risks of the study product ALT001, thereby providing scientific, detailed and reliable evidence-based medical data to optimize clinical treatment guidelines and formulate individualized treatment regimens for knee osteoarthritis.

This clinical trial is conducted in response to the urgent clinical need for safe and effective interventions in the treatment of knee osteoarthritis. In accordance with the principles of evidence-based medicine, a rigorous controlled study protocol has been designed. Through standardized trial procedures and a unified evaluation system, this study will systematically and comprehensively assess the clinical efficacy of ALT001, manufactured by Darwin Starting Point (Hubei) Biopharmaceutical Co., Ltd., in patients with knee osteoarthritis. The trial will focus on core efficacy endpoints including the relief of pain intensity, improvement of joint motor function and enhancement of patients' quality of life. Meanwhile, it will strictly monitor key safety indicators such as the occurrence of various adverse events following medication administration, as well as the severity and duration of adverse reactions, and conduct a multi-dimensional and multi-level comprehensive assessment. The aim is to clarify the clinical benefit profile and safety risks of the investigational product ALT001, and to provide scientific, detailed and reliable evidence-based medical data to support the optimization of clinical treatment guidelines and the formulation of individualized treatment regimens for knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50 to 75 years old (inclusive), gender unrestricted;
2. Body Mass Index (BMI) within the range of 18 ≤ BMI ≤ 35;
3. Meets the diagnostic criteria for osteoarthritis (OA) in Chinese Guidelines for the Diagnosis and Treatment of Osteoarthritis (2021 Edition) [1]. A diagnosis of knee osteoarthritis can be made if criterion ① plus any 2 of criteria ②, ③, ④, ⑤ are satisfied:

   ① Recurrent knee pain within the past 1 month;

   ② X-ray (standing or weight-bearing position) shows narrowed joint space, subchondral bone sclerosis and/or cystic changes, and osteophyte formation at the joint margin;

   ③ Aged ≥ 50 years;

   ④ Morning stiffness duration ≤ 30 minutes;

   ⑤ Crepitus (sensation or sound) during joint movement;
4. Kellgren-Lawrence grade of Grade Ⅰ to Ⅲ for at least one knee joint on anteroposterior and lateral (stress) X-ray of bilateral knee joints within 6 months;
5. A score of 4 to 8 points (inclusive) for pain on flat ground walking or stair climbing in the WOMAC Pain Score of at least one knee joint;
6. For participants who have been taking glucosamine or diacerein-containing drugs before the screening period, the dosage must be kept stable throughout the entire clinical trial;
7. Discontinued all analgesic drugs for more than 2 weeks before the screening period, and agreed not to use any other analgesic drugs except rescue medication throughout the entire study;
8. Willing to cooperate with the clinical trial and able to sign the informed consent form.

Exclusion Criteria:

1. With other diseases that cause knee pain and dysfunction (e.g., autoimmune arthritis, infectious arthritis, gouty arthritis, knee joint tumors, etc.);
2. With pain in other body parts exceeding knee pain, which may interfere with the assessment of the knee joint;
3. With significantly narrowed joint space or bony ankylosis due to bone bridge formation between joints;
4. With lower extremity pain caused by lumbar spinal stenosis or lumbar disc herniation;
5. With systemic infection or severe local infection;
6. With clinically significant abnormalities in any item of the four infectious disease screening tests;
7. With a history of knee joint surgery, open trauma within 1 year, or intra-articular injection, radiotherapy, or arthroscopy within 6 months;
8. With intra-articular corticosteroid block therapy for the knee joint or long-term (continuous ≥2 weeks) use of corticosteroids or immunosuppressants within 6 months;
9. With a history of taking Chinese herbal decoctions or proprietary Chinese medicines for knee pain within 1 month;
10. With physical therapy or topical medication (e.g., electromagnetic therapy, cupping, acupuncture, plasters, fumigation, etc.) on the knee joint within 1 week;
11. With severe diseases of the heart, brain, liver, kidney, hematologic, endocrine, or immune systems (e.g., AST/ALT or creatinine ≥2.0×ULN, glycosylated hemoglobin ≥8%, hemophilia, etc.);
12. With malignant tumors;
13. Planning to undergo elective knee joint surgery during the study period;
14. With obvious knee joint effusion (significant joint swelling or bulging) or severe venous/lymphatic stasis of the lower extremities;
15. Requiring long-term use of warfarin or other anticoagulants (except for a stable daily dose of aspirin ≤100 mg and/or clopidogrel);
16. With consciousness disturbance or mental illness, unable to complete self-assessment;
17. With a history of drug abuse or alcoholism;
18. With a history of allergy to the raw materials of the study product and control product, or atopic diathesis (previous allergy to protein-based drugs or food);
19. With a positive pregnancy test, pregnant/lactating women, those with recent childbearing plans, or those unable to take reliable contraceptive measures during the study;
20. Having participated in other clinical trials of drugs, biological agents, or medical products within 3 months;
21. Other circumstances deemed inappropriate for participation in this clinical trial by the investigator.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the WOMAC Pain Score of the target knee joint at 24 weeks (14 weeks after the last injection) compared with the baseline. | 24 weeks (14 weeks after the last injection)
  The WOMAC Index (Western Ontario and McMaster Universities Osteoarthritis Index) is a commonly used assessment tool for evaluating symptom severity and joint function in patients with knee joint disorders [6]. It comprises three dimensions: pain, stiffness, and physical function. Through the assessment of these three dimensions, the degree of pain, joint mobility, and difficulty in performing daily activities in patients' daily lives can be objectively evaluated. The WOMAC score is a composite rating of the patient's subjective experience within the 48 hours prior to each assessment.
  WOMAC Pain Score includes five items: pain when walking on a flat surface, climbing up or down stairs, pain at night, pain when sitting or lying down, and pain when standing upright. For detailed scoring criteria, see Annex 1. During the treatment period and the final follow-up period, the pain assessment is based on the patient's experience within the 48 hours prior to the current visit.
Changes in the levels of inflammatory factors IL-1β, IL-6, and TNF-α in the synovial fluid of the target knee joint during treatment and at 14 weeks post-treatment compared with the baseline. | 14 weeks
  IL-1β, IL-6, and TNF-α, the three cytokines, can promote the production of other inflammatory factors by activating the NF-κB and MAPK signaling pathways, thereby exacerbating the degree of inflammatory response. Although this interaction can trigger a more robust immune response, it may also induce chronic inflammation and tissue damage. The levels of IL-1β, IL-6, and TNF-α serve as important predictive markers for monitoring the disease progression of osteoarthritis (OA). (For patients from whom synovial fluid cannot be aspirated, irrigate the joint cavity with 5 ml of sterile water for injection first before aspiration; the entire procedure must be performed under strict aseptic conditions.)

SECONDARY OUTCOMES:
Changes in the WOMAC Physical Function Score of the target knee joint at 2, 4, 6, 8, 10, 12, 18 (non-mandatory) and 24 weeks compared with the baseline. | 2, 4, 6, 8, 10, 12, 18(non-mandatory)
  WOMAC Physical Function: It includes 17 items: climbing up stairs, climbing down stairs, rising from a seated position, walking on a flat surface, getting in/out of a car, going shopping, putting on socks, rising from a bed, taking off socks, lying in bed, getting in/out of a bathtub, sitting down, rising from a toilet, doing heavy housework, and doing light housework.
Changes in the WOMAC Total Score of the target knee joint at 2, 4, 6, 8, 10, 12, 18 (non-mandatory) and 24 weeks compared with the baseline. | 2, 4, 6, 8, 10, 12, 18 (non-mandatory) and 24 weeks
  The sum of the pain, stiffness and physical function scores in the WOMAC Index.
Changes in the VAS Pain Score of the target knee joint at 2, 4, 6, 8, 10, 12, 18 (non-mandatory) and 24 weeks compared with the baseline. | 2, 4, 6, 8, 10, 12, 18 (non-mandatory) and 24 weeks
  Based on the patient's subjective pain rating.

IPD SHARING:
Plan to Share IPD: Yes
Wherever possible, appropriately anonymised datasets from the sponsor-funded research will be made available for further analysis,Publications related to this study may be requested for access via the email address: xiaodongguo@hust.edu.cn.
Supporting Information: Study Protocol, ICF
Time Frame: After the project finished，publications on this study will be available from PubMed.
Access Criteria: Relevant data may be requested via xiaodongguo@hust.edu.cn.